CLINICAL TRIAL: NCT01504178
Title: Evaluation of the Role of the Noradrenergic System in Pain Perception in Parkinson's Disease
Acronym: DOULOX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: French Parkinson Association (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 09 303 03
Record Dates: First submitted 2011-12-30; First posted 2012-01-05 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Parkinson's Disease
Keywords: Noradrenergic system and pain in Parkinson's disease
MeSH Terms: conditions — Parkinson Disease | interventions — Duloxetine Hydrochloride; Levodopa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- duloxetine (Experimental): The first group (12 patients) will receive, after 28 days of duloxetine treatment, one duloxetine dose, an injection of apomorphine and a placebo of L-Dopa.
  Interventions: Drug: duloxetine; Drug: injection of apomorphine; Drug: injection of placebo of L-Dopa
- positive control (L-Dopa) (Placebo Comparator): The second group (12 patients) will receive, after 28 days of placebo treatment, one placebo dose of duloxetine, an injection of apomorphine and injection of placebo of L-Dopa.
  Interventions: Drug: placebo of duloxetine; Drug: injection of apomorphine; Drug: injection of placebo of L-Dopa
- negative control (Placebo Comparator): The third group will receive, after 28 days of placebo treatment, one placebo of duloxetine, an injection of placebo of apomorphine and a dose of L-Dopa.
  Interventions: Drug: placebo of duloxetine; Drug: injection of placebo of apomorphine; Drug: L-Dopa

INTERVENTIONS:
Drug: duloxetine — administration during 28 days
  Arms: duloxetine
Drug: placebo of duloxetine — administration during 28 days
  Arms: negative control; positive control (L-Dopa)
Drug: injection of apomorphine — injection performed at D28
  Arms: duloxetine; positive control (L-Dopa)
Drug: injection of placebo of apomorphine — performed at D28
  Arms: negative control
Drug: L-Dopa — performed at D28
  Other Names: injection of L-dopa
  Arms: negative control
Drug: injection of placebo of L-Dopa — performed at D28
  Arms: duloxetine; positive control (L-Dopa)

SUMMARY:
Patients suffering from Parkinson's disease (PD) frequently experienced painful sensations that could be, in part, due to a central modification of nociception mechanisms. Previous studies have shown that pain perception was altered in Parkinson's disease (subjective and objective pain thresholds and pain-induced cerebral activity) and that administration of L-Dopa normalized this alteration. In the central nervous system, L-Dopa is converted in dopamine and in norepinephrine. Apomorphine (a dopamine agonist) has no effect on pain threshold and pain-induced cerebral activity. Therefore the noradrenergic system could be involved in pain alteration in PD.

To assess the role of noradrenergic system in pain in patients with PD, we chose duloxetine (norepinephrine and serotonin reuptake inhibitor)because a recent study had shown that duloxetine allowed an improvement of pain clinical scores (pain questionnaires) in patients with PD.

36 patients will be enrolled in this study. We supposed that a chronic intake of duloxetine increase the pain perception level compare to the placebo. This increase would be the same than those observed with L-Dopa.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinical diagnosis of Parkinson's disease according to the criteria of the UKPDSBB
* Parkinson's disease patients with a score ≤ 3 on the Hoehn and Yahr scale
* Patients treated with dopaminergic antiparkinsonian drugs (L-Dopa, dopamine agonists, ICOMT…)
* Patients affiliated to a social protection program
* Women with efficacy contraception

Exclusion Criteria:

* Patients suffering from another pathology causing chronic pain (rheumatic disease, traumatic or orthopedic pathologies…)
* Parkinson's disease patients with a score > 3 on the Hoehn and Yahr scale
* Depressed patients (MADRS score < 16)
* Patients suffering from a cancer
* Patients under tutelage, curatella or law protection
* Patients with a complete contraindication against apomorphine injections or duloxetine administration (selective serotonin reuptake inhibitor and monoamine oxydase inhibitors)
* Patients without any control of their arterial hypertension
* Patients with a neuroleptic treatment
* Pregnant women

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2011-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Subjective pain threshold determined using thermal stimulations (thermotest) with the method of levels | One month
  Before duloxetine intake and after one month of chronic duloxetine intake

SECONDARY OUTCOMES:
Objective pain threshold determined recording the nociceptive reflex of flexion | One month
  Before duloxetine intake and after one month of chronic duloxetine intake
Clinical evaluation of the severity of the motor handicap of patients using the Unified Parkinson's Disease Rating Scale (UPDRS III) | One month
  Before duloxetine intake and after one month of chronic duloxetine intake

CONTACTS AND LOCATIONS:
Overall Officials: Christine Brefel-Courbon, MD, Principal Investigator — Purpan hospital, Toulouse
Locations (1):
- CIC, Purpan Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: Undecided